CLINICAL TRIAL: NCT05651217
Title: A Multicenter, Prospective, Randomized Controlled Clinical Study to Evaluate the Safety and Effectiveness of Disposable Sterile Urinary Catheter
Brief Title: Clinical Study on Disposable Sterile Urinary Catheter
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The production of control group products is stopped, and the control group products cannot be obtained
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B201703
Record Dates: First submitted 2022-12-01; First posted 2022-12-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Urinary Catheters; Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): Patients in this group used the disposable urinary catheter
  Interventions: Device: disposable urinary catheter
- control group (Active Comparator): Patients in this group used super smooth antibacterial urinary catheter
  Interventions: Device: super smooth antibacterial urinary catheter

INTERVENTIONS:
Device: disposable urinary catheter — The trial group was intervened with disposable sterile urinary catheter. The model of the trial group includes two chamber type (Fr8, Fr10, Fr12, Fr14, Fr16, Fr18, Fr20, Fr22, Fr24) and three chamber type (Fr16, Fr18, Fr20, Fr22, Fr24).
  Arms: trial group
Device: super smooth antibacterial urinary catheter — the control group was intervened with ultra smooth antibacterial catheter. The control group models include single chamber (6Fr, 8Fr, 10Fr, 12Fr, 14Fr, 16Fr, 18Fr, 20Fr, 22Fr, 24Fr), double chamber (6Fr, 8Fr, 10Fr, 12Fr, 14Fr, 16Fr, 18Fr, 20Fr, 22Fr, 24Fr, 26Fr, 28Fr, 30Fr), and three chamber (16Fr, 18Fr, 20Fr, 22Fr, 24Fr, 26Fr)
  Arms: control group

SUMMARY:
This study is a multicenter, randomized controlled study, with the urinary tract infection rate at the time of catheter insertion for 1 week as the primary end point. By comparing the clinical safety and effectiveness of two kinds of urethral catheters, to evaluate the clinical application effect of one kind of urethral catheters.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year old patients;
* Retained catheter ≥ 7 days;
* Patients who were conscious and had good communication skills and volunteered to participate in the study.

Exclusion Criteria:

* Pregnant and lactating female patients;
* Diabetes patients;
* Patients allergic to sulfadiazine, silica gel and stainless steel;
* Urethral malformation, acute urethral injury, prostate disease, intermittent catheterization, suprapubic cystostomy and other patients who are not suitable for catheterization;
* Patients who have used urinary catheters for a long time or had catheters retained within one week;
* Patients who are participating in other clinical trials that interfere with this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection rate | one week
  In accordance with the "Diagnostic Criteria for Catheter associated Urinary Tract Infection" in the "Technical Guidelines for the Prevention and Control of Catheter associated Urinary Tract Infection (Trial)" formulated and issued by the Ministry of Health in 2011. Although the patient has no symptoms, he or she has endoscopic examination or catheterization within one week. If the number of Gram positive cocci colonies in urine culture ≥ 10 has 4 cfu/ml, and the number of Gram negative bacilli colonies ≥ 10 has 5 cfu/ml, he or she should be diagnosed as asymptomatic bacteriuria. If the patient has urinary tract irritation symptoms such as frequent urination, urgent urination, and painful urination, or has lower abdominal tenderness, renal area percussion pain, with or without fever (>38.0 ℃), it is symptomatic bacteriuria.

SECONDARY OUTCOMES:
Success rate of catheterization | 10 minutes after catheterization
  The success of catheterization is based on the evaluation of each instrument, which can be placed at the catheterization site as expected and catheterization can be carried out smoothly.
level of urethral irritation | 10 minutes after catheterization
  Level 0, no discomfort at all; Grade I, slight discomfort, but tolerable; Grade II, moderate discomfort, intolerable, urgency of urination, urethral pain, abdominal distension; Grade III, severe discomfort, extremely intolerable, obvious distension of lower abdomen, urethral pain, urgency of urination, and the desire to pull out the catheter, accompanied by restlessness, increased heart rate, and elevated blood pressure.
level of urethral irritation | 72 hours
  Level 0, no discomfort at all; Grade I, slight discomfort, but tolerable; Grade II, moderate discomfort, intolerable, urgency of urination, urethral pain, abdominal distension; Grade III, severe discomfort, extremely intolerable, obvious distension of lower abdomen, urethral pain, urgency of urination, and the desire to pull out the catheter, accompanied by restlessness, increased heart rate, and elevated blood pressure.
level of urethral irritation | one week
  Level 0, no discomfort at all; Grade I, slight discomfort, but tolerable; Grade II, moderate discomfort, intolerable, urgency of urination, urethral pain, abdominal distension; Grade III, severe discomfort, extremely intolerable, obvious distension of lower abdomen, urethral pain, urgency of urination, and the desire to pull out the catheter, accompanied by restlessness, increased heart rate, and elevated blood pressure.
Incidence of device related adverse events | 72 hours
  The safety of clinical use of the device was evaluated based on the incidence of adverse events related to the device that occurred after the subject placed the tube. Including: balloon leakage, rupture, catheter self falling off, difficulty in pulling out catheter, catheter blockage, urine retention, urine leakage, hematuria, urethral injury, etc; It can be judged according to clinical experience, and imaging methods can be used when necessary.
Incidence of device related adverse events | one week
  The safety of clinical use of the device was evaluated based on the incidence of adverse events related to the device that occurred after the subject placed the tube. Including: balloon leakage, rupture, catheter self falling off, difficulty in pulling out catheter, catheter blockage, urine retention, urine leakage, hematuria, urethral injury, etc; It can be judged according to clinical experience, and imaging methods can be used when necessary.
time of catheter duration | one week
  Time from insertion to removal of catheter
rating of operation convenience | 10 minutes after catheterization
  Including excellent: very convenient, good: relatively convenient, poor: poor convenience
rate of packaging integrity | 10 minutes after catheterization
rate of device defect rate | 10 minutes after catheterization
  The package is damaged, the balloon cannot be inflated, and the balloon leaks or breaks

CONTACTS AND LOCATIONS:
Locations (1):
- Liaoning Cancer Hospital & institute, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No